CLINICAL TRIAL: NCT00402233
Title: A Randomized, Double-blind, Active (Pramipexole 0.5 mg Tid) and Placebo Controlled, Efficacy Study of Pramipexole Given 0.5 mg and 0.75 mg Bid Over a 12-week Treatment Phase in Early Parkinson's Disease Patients (PramiBID)
Brief Title: A Randomized, Double-blind, Active (Pramipexole 0.5 mg Tid) and Placebo Controlled, Study of Pramipexole Given 0.5 mg and 0.75 mg Bid Over 12-week Treatment in Early Parkinson's Disease (PD) Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 248.622; PramiBID
Record Dates: First submitted 2006-11-19; First posted 2006-11-22 (Estimated); Results first posted 2010-01-13 (Estimated); Last update posted 2014-05-16 (Estimated); Status verified 2014-05

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Pramipexole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- Placebo (Other)
  Interventions: Drug: Placebo
- Pramipexole 0.5 mg Tid (Other): Pramipexole 0.5 mg tid (three times a day)
  Interventions: Drug: Pramipexole
- Pramipexole 0.5 mg Bid (Other): Pramipexole 0.5 mg bid (bis in die (two times a day))
  Interventions: Drug: Pramipexole
- Pramipexole 0.75 mg Bid (Other): Pramipexole 0.75 mg bid (bis in die (two times a day))
  Interventions: Drug: Pramipexole

INTERVENTIONS:
Drug: Pramipexole
  Arms: Pramipexole 0.5 mg Bid; Pramipexole 0.5 mg Tid; Pramipexole 0.75 mg Bid
Drug: Placebo
  Arms: Placebo

SUMMARY:
Primary objective: to assess the efficacy of pramipexole given two times daily compared to placebo.

Secondary objectives: to assess the effects of pramipexole on mood, cognition, fatigue, impulse control, daytime sleepiness and nighttime sleep compared to placebo; to compare the tolerability among the treatment groups over 12 weeks

ELIGIBILITY:
Inclusion Criteria:

Potential subjects must meet all of the following inclusion criteria to be eligible for enrollment into this study:

1. Must be willing and able to give informed consent.
2. Must be over 30 years of age at Baseline.
3. Must have idiopathic Parkinson's disease of less than 7 years duration since diagnosis, characterized by 2 of the following 3 cardinal signs (signs need to be asymmetric): resting tremor, bradykinesia and rigidity.
4. Must have a Modified Hoehn and Yahr stage <3.
5. Should be able to safely tolerate placebo for up to 12 weeks after Baseline.
6. Must have a negative urine pregnancy test at the Screening Visit and use an adequate contraceptive method throughout the study if a woman of child-bearing potential. Women who are surgically sterile (hysterectomy or tubal ligation) or whose last menstruation was 12 months or more prior to the Screening Visit are considered to be of non-child-bearing potential. Acceptable forms of contraception include oral, implanted, or injected contraceptives intrauterine devices in place for at least 3 months estrogen patch and adequate barrier methods in conjunction with spermicide. Abstinence is considered an acceptable contraceptive regimen.
7. Must be willing and able to comply with trial procedures. They must be sufficiently proficient in English to understand and complete study instruments.

Exclusion Criteria:

Individuals with any of the following characteristics will not be eligible for entry into this study:

1. Signs or symptoms suggesting other parkinsonian syndromes.
2. Use of medications that may cause secondary parkinsonism, including but not limited to: neuroleptics, metaclopramide, alphamethyldopa, flunarizine, methylphenidate, cinnarizine, reserpine, or amphetamines in the last 6 months prior to Baseline Visit.
3. Use of dopaminergic medications within the last 3 months or for longer than 6 months prior to Baseline Visit.
4. Presence of dementia by Diagnostic and Statistical Manual of Mental Disorders IV criteria (R06-1340) or a Mini Mental State Examination (R96-2656) (Appendix 10.1) score less than 26 at Screening Visit.
5. Presence of major depression, as determined by medical history.
6. Active epilepsy (i.e., occurrence of a seizure) within the past year prior to Baseline Visit.
7. Electro Convulsive Therapy in previous 90 days prior to Baseline Visit.
8. Myocardial infarction within previous 6 months prior to Baseline Visit.
9. Third degree atrioventricular block or sick sinus syndrome.
10. Congestive heart failure Class III or IV by New York Heart Association classification.
11. Symptomatic orthostatic hypotension at Screening Visit.
12. Stereotaxic brain surgery.
13. Clinically significant liver disease.
14. Clinically significant renal disease.
15. Any other clinically significant medical or psychiatric condition (e.g., angina, active neoplasm) that in the judgment of the investigator would interfere with the subjects ability to participate in the study or would jeopardize safe conduct of the study.
16. Breastfeeding.
17. Known hypersensitivity or intolerability to pramipexole.
18. Participating in other drug studies or receiving other experimental medications within 30 days of Baseline Visit.
19. History of drug or alcohol dependency within 6 months of baseline visit.

Min Age: 31 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Actual)
Dates: Start 2006-11; Primary Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (39):
- United States (39):
  - 248.622.170 Boehringer Ingelheim Investigational Site, Phoenix, Arizona
  - 248.622.112 Boehringer Ingelheim Investigational Site, Little Rock, Arkansas
  - 248.622.69 Boehringer Ingelheim Investigational Site, Fountain Valley, California
  - 248.622.198 Boehringer Ingelheim Investigational Site, La Jolla, California
  - 248.622.111 Boehringer Ingelheim Investigational Site, Oxnard, California
  - 248.622.61 Boehringer Ingelheim Investigational Site, Sacramento, California
  - 248.622.23 Boehringer Ingelheim Investigational Site, San Diego, California
  - 248.622.73 Boehringer Ingelheim Investigational Site, San Francisco, California
  - 248.622.108 Boehringer Ingelheim Investigational Site, Denver, Colorado
  - 248.622.190 Boehringer Ingelheim Investigational Site, Danbury, Connecticut
  - 248.622.215 Boehringer Ingelheim Investigational Site, Manchester, Connecticut
  - 248.622.196 Boehringer Ingelheim Investigational Site, Boca Raton, Florida
  - 248.622.14 Boehringer Ingelheim Investigational Site, Miami, Florida
  - 248.622.149 Boehringer Ingelheim Investigational Site, Weston, Florida
  - 248.622.139 Boehringer Ingelheim Investigational Site, Honolulu, Hawaii
  - 248.622.5 Boehringer Ingelheim Investigational Site, Chicago, Illinois
  - 248.622.138 Boehringer Ingelheim Investigational Site, Springfield, Illinois
  - 248.622.87 Boehringer Ingelheim Investigational Site, Louisville, Kentucky
  - 248.622.207 Boehringer Ingelheim Investigational Site, New Orleans, Louisiana
  - 248.622.132 Boehringer Ingelheim Investigational Site, Shreveport, Louisiana
  - 248.622.17 Boehringer Ingelheim Investigational Site, Boston, Massachusetts
  - 248.622.40 Boehringer Ingelheim Investigational Site, Boston, Massachusetts
  - 248.622.76 Boehringer Ingelheim Investigational Site, Boston, Massachusetts
  - 248.622.186 Boehringer Ingelheim Investigational Site, East Lansing, Michigan
  - 248.622.77 Boehringer Ingelheim Investigational Site, Omaha, Nebraska
  - 248.622.155 Boehringer Ingelheim Investigational Site, Lebanon, New Hampshire
  - 248.622.135 Boehringer Ingelheim Investigational Site, Brooklyn, New York
  - 248.622.216 Boehringer Ingelheim Investigational Site, Kingston, New York
  - 248.622.202 Boehringer Ingelheim Investigational Site, New York, New York
  - 248.622.86 Boehringer Ingelheim Investigational Site, New York, New York
  - 248.622.1 Boehringer Ingelheim Investigational Site, Rochester, New York
  - 248.622.89 Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - 248.622.20 Boehringer Ingelheim Investigational Site, Columbus, Ohio
  - 248.622.169 Boehringer Ingelheim Investigational Site, Hershey, Pennsylvania
  - 248.622.18 Boehringer Ingelheim Investigational Site, Philadelphia, Pennsylvania
  - 248.622.199 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 248.622.7 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 248.622.213 Boehringer Ingelheim Investigational Site, Spokane, Washington
  - 248.622.104 Boehringer Ingelheim Investigational Site, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were 312 patients enrolled and 311 patients entered
Groups:
- Placebo: matching tablet
- Mirapex (Pramipexole 0.5 mg Tid): Week 1: Pramipexole 0.125 mg tid, Week 2: Pramipexole 0.25 mg tid, Week 3: Pramipexole 0.5 mg tid, Week 4 to Week 12: Pramipexole 0.5 mg tid. After the initial 4 week titration period, each dosage group will maintain the specified dosage for an additional 8 weeks, to complete the 12 week double-blind period.
- Mirapex (Pramipexole 0.5 mg Bid): Week 1: Pramipexole 0.125 mg bid, Week 2: Pramipexole 0.25 mg bid, Week 3: Pramipexole 0.5 mg bid, Week 4 to Week 12: Pramipexole 0.5 mg bid. After the initial 4 week titration period, each dosage group will maintain the specified dosage for an additional 8 weeks, to complete the 12 week double-blind period.
- Mirapex (Pramipexole 0.75 mg Bid): Week 1: Pramipexole 0.125 mg bid, Week 2: Pramipexole 0.25 mg bid, Week 3: Pramipexole 0.5 mg bid, Week 4 to Week 12: Pramipexole 0.75 mg bid. After the initial 4 week titration period, each dosage group will maintain the specified dosage for an additional 8 weeks, to complete the 12 week double-blind period.
Period: Overall Study
Arm/Group | Placebo | Mirapex (Pramipexole 0.5 mg Tid) | Mirapex (Pramipexole 0.5 mg Bid) | Mirapex (Pramipexole 0.75 mg Bid)
Started | 77 | 80 | 81 | 73
Completed | 72 | 70 | 70 | 62
Not Completed | 5 | 10 | 11 | 11
Not completed — Adverse Event | 1 | 7 | 9 | 9
Not completed — Protocol Violation | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 2 | 2
Not completed — Worsening of disease under study | 2 | 0 | 0 | 0
Not completed — Worsening of other pre-existing disease | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Mirapex (Pramipexole 0.5 mg Tid) | Mirapex (Pramipexole 0.5 mg Bid) | Mirapex (Pramipexole 0.75 mg Bid) | Total
Number analyzed (Participants) | 77 | 80 | 81 | 73 | 311
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.7 (11) | 63.7 (9.8) | 61.6 (10.2) | 63.1 (9.9) | 62.3 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 23 | 30 | 32 | 104
  Male | 58 | 57 | 51 | 41 | 207

OUTCOME MEASURES:

1. Primary Outcome: Unified Parkinson's Disease Rating Scale (UPDRS) Total Score
Description: Total score ranges from zero (best) to 176 (worst), as the sum of Parts I (Mental questions), II (Activity of Daily Living questions), and III (Motor examination)
Time Frame: From baseline to week 12
Population: Treated set
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Mirapex (Pramipexole 0.5 mg Tid) | Mirapex (Pramipexole 0.5 mg Bid) | Mirapex (Pramipexole 0.75 mg Bid)
Number analyzed (Participants) | 77 | 80 | 81 | 73
units on a scale
  UPDRS at baseline | 28.97 (11.82) | 27.66 (10.72) | 27.21 (11.76) | 27.77 (9.18)
  UPDRS at week 12 | 28.19 (12.94) | 22.92 (10.44) | 22.96 (11.94) | 22.65 (10.82)
Statistical Analysis 1: Comparison: Placebo vs Mirapex (Pramipexole 0.5 mg Tid); Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -4.4, 95% CI [-6.53 to -2.26]
Statistical Analysis 2: Comparison: Placebo vs Mirapex (Pramipexole 0.5 mg Bid); Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -4.41, 95% CI [-6.54 to -2.28]
Statistical Analysis 3: Comparison: Placebo vs Mirapex (Pramipexole 0.75 mg Bid); Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -4.72, 95% CI [-6.91 to -2.52]

2. Secondary Outcome: Modified Hoehn and Yahr Stage
Description: Score ranges from best 0 (no signs of disease) to worst 5 (wheelchair bound or bedridden unless aided)
Time Frame: From baseline to week 12
Population: Treated set
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Mirapex (Pramipexole 0.5 mg Tid) | Mirapex (Pramipexole 0.5 mg Bid) | Mirapex (Pramipexole 0.75 mg Bid)
Number analyzed (Participants) | 77 | 80 | 81 | 73
units on a scale
  Modified Hoehn and Yahr Stage at baseline | 1.81 (0.48) | 1.74 (0.5) | 1.72 (0.5) | 1.73 (0.51)
  Modified Hoehn and Yahr Stage at week 12 | 1.74 (0.54) | 1.68 (0.52) | 1.69 (0.52) | 1.62 (0.56)
Statistical Analysis 1: Comparison: Placebo vs Mirapex (Pramipexole 0.5 mg Tid); Test type: Superiority or Other; Regression, Logistic; Odds Ratio (OR) = 0.893, 95% CI [0.431 to 1.849]
Statistical Analysis 2: Comparison: Placebo vs Mirapex (Pramipexole 0.5 mg Bid); Test type: Superiority or Other; Regression, Logistic; Odds Ratio (OR) = 0.885, 95% CI [0.424 to 1.845]
Statistical Analysis 3: Comparison: Placebo vs Mirapex (Pramipexole 0.75 mg Bid); Test type: Superiority or Other; Regression, Logistic; Odds Ratio (OR) = 0.687, 95% CI [0.317 to 1.492]

3. Secondary Outcome: Epworth Sleepiness Scale
Description: Total score ranges from zero (best) to 24 (worst); scale has 8 items, each rated from zero (no chance of dozing) to 3 (high chance of dozing)
Time Frame: From baseline to week 12
Population: Treated set
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Mirapex (Pramipexole 0.5 mg Tid) | Mirapex (Pramipexole 0.5 mg Bid) | Mirapex (Pramipexole 0.75 mg Bid)
Number analyzed (Participants) | 77 | 80 | 81 | 73
units on a scale
  Epworth Sleepiness Scale at baseline | 5.29 (3.47) | 5.8 (3.66) | 5.78 (3.74) | 6.34 (4.35)
  Epworth Sleepiness Scale at week 12 | 5.09 (3.33) | 6.58 (3.62) | 6.44 (4.21) | 7.52 (5.03)
Statistical Analysis 1: Comparison: Placebo vs Mirapex (Pramipexole 0.5 mg Tid); Test type: Superiority or Other; p = 0.014, ANCOVA; Mean Difference (Final Values) = 1.14, 95% CI [0.23 to 2.04]
Statistical Analysis 2: Comparison: Placebo vs Mirapex (Pramipexole 0.5 mg Bid); Test type: Superiority or Other; p = 0.03, ANCOVA; Mean Difference (Final Values) = 1, 95% CI [0.094 to 1.9]
Statistical Analysis 3: Comparison: Placebo vs Mirapex (Pramipexole 0.75 mg Bid); Test type: Superiority or Other; p = 0.0019, ANCOVA; Mean Difference (Final Values) = 1.49, 95% CI [0.56 to 2.43]

4. Secondary Outcome: Beck Depression Inventory II
Description: Total score ranges from zero (best) to 63 (worst); scale has 21 items, each rated from zero (absent) to 3 (severe)
Time Frame: From baseline to week 12
Population: Treated set
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Mirapex (Pramipexole 0.5 mg Tid) | Mirapex (Pramipexole 0.5 mg Bid) | Mirapex (Pramipexole 0.75 mg Bid)
Number analyzed (Participants) | 77 | 80 | 81 | 73
units on a scale
  Beck Depression Inventory II at baseline | 6.05 (6.01) | 6.66 (5.36) | 6.96 (5.14) | 7.4 (5.87)
  Beck Depression Inventory II at week 12 | 5.92 (5.83) | 5.70 (5.14) | 5.97 (5.14) | 6.54 (5.19)
Statistical Analysis 1: Comparison: Placebo vs Mirapex (Pramipexole 0.5 mg Tid); Test type: Superiority or Other; p = 0.39, ANCOVA; Mean Difference (Final Values) = -0.55, 95% CI [-1.82 to 0.71]
Statistical Analysis 2: Comparison: Placebo vs Mirapex (Pramipexole 0.5 mg Bid); Test type: Superiority or Other; p = 0.37, ANCOVA; Mean Difference (Final Values) = -0.57, 95% CI [-1.84 to 0.69]
Statistical Analysis 3: Comparison: Placebo vs Mirapex (Pramipexole 0.75 mg Bid); Test type: Superiority or Other; p = 0.48, ANCOVA; Mean Difference (Final Values) = -0.47, 95% CI [-1.78 to 0.84]

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Placebo | Mirapex (Pramipexole 0.5 mg Bid) | Mirapex (Pramipexole 0.75 mg Bid) | Mirapex (Pramipexole 0.5 mg Tid)
Serious Adverse Events (participants affected / at risk) | 0/77 | 0/81 | 2/73 | 1/80
Other Adverse Events (participants affected / at risk) | 27/77 | 42/81 | 37/73 | 43/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=77) | Mirapex (Pramipexole 0.5 mg Bid) (N=81) | Mirapex (Pramipexole 0.75 mg Bid) (N=73) | Mirapex (Pramipexole 0.5 mg Tid) (N=80)
Coronary Artery Disease (Cardiac disorders) | 0 | 0 | 1 | 0
Cerebral Infarction, Hemiparesis (Nervous system disorders) | 0 | 0 | 1 | 0
ileus (patient stopped drugs 2 days prior) (Gastrointestinal disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=77) | Mirapex (Pramipexole 0.5 mg Bid) (N=81) | Mirapex (Pramipexole 0.75 mg Bid) (N=73) | Mirapex (Pramipexole 0.5 mg Tid) (N=80)
somnolence (Nervous system disorders) | 4 | 14 | 16 | 20
dizziness (Nervous system disorders) | 7 | 9 | 5 | 9
headache (Nervous system disorders) | 8 | 7 | 6 | 4
tremor (Nervous system disorders) | 4 | 1 | 3 | 0
nausea (Gastrointestinal disorders) | 7 | 18 | 11 | 15
constipation (Gastrointestinal disorders) | 2 | 8 | 7 | 5
insomnia (Psychiatric disorders) | 4 | 3 | 9 | 5
abnormal dreams (Psychiatric disorders) | 3 | 3 | 2 | 5
fatigue (General disorders) | 3 | 6 | 7 | 4
oedema peripheral (General disorders) | 0 | 2 | 4 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.